CLINICAL TRIAL: NCT04426214
Title: Neuromodulation and Cognitive Training for Substance Use Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSYCH-2020-28848
Record Dates: First submitted 2020-05-29; First posted 2020-06-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Stimulant Use; Alcohol Use Disorder
Keywords: tDCS; Cognitive Training; Plasticity
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS (Experimental)
  Interventions: Device: tDCS; Behavioral: Cognitive Training
- Sham tDCS (Placebo Comparator)
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Device: tDCS — We will apply tDCS in combination with cognitive training. All participants receive cognitive training, and will be randomized to receive either active or sham tDCS
  Arms: Active tDCS
Behavioral: Cognitive Training — cognitive training on computer

SUMMARY:
The relapsing nature of substance use disorder is a major obstacle to successful treatment. About 70% of those entering treatment will relapse within one year. To improve treatment outcome, new interventions targeting the underlying brain biomarkers of relapse vulnerability hold significant promise in reducing this critical public health problem. This study is testing a new intervention, namely tDCS-Augmented Cognitive Training, to engage these brain biomarkers to improve cognition and improve treatment outcomes.

DETAILED DESCRIPTION:
The relapsing nature of substance use disorder is a major obstacle to successful treatment. About 70% of those entering treatment will relapse within one year. To improve treatment outcome, new interventions targeting the underlying brain biomarkers of relapse vulnerability hold significant promise in reducing this critical public health problem.

Preliminary Data: Using resting functional magnetic resonance imaging (fMRI) we have identified brain biomarkers that support long-term abstinence. Our cross-sectional and longitudinal findings provide evidence that higher FC, particularly between NAcc and DLPFC, is a potential brain biomarker that supports abstinence. Long-term abstinent alcoholics (7 years of abstinence) have higher resting FC between NAcc and DLPFC when compared to controls. Short-term abstinent alcoholics (11 weeks of abstinence) have intermediate FC (lower than long-term abstinent alcoholics and higher than controls) (Camchong, Stenger, & Fein, 2013b, 2013c). Further, lower FC between NAcc and DLPFC at 11 weeks of abstinence can be a predictor of subsequent relapse (with 74% accuracy) (Camchong, Stenger, & Fein, 2013a). Moreover, in a pilot longitudinal FC study examining resting FC of NAcc at 5 and 13 weeks of abstinence in individuals with stimulant use disorder, we found that FC between NAcc and DLPFC decreased from 5 to 13 weeks of abstinence in subsequent relapsers, while it increased in subsequent abstainers (Camchong et al., 2014). Based on the above, we believe that long-term abstinence is supported by a compensatory mechanism that mediates proper executive function over reward (mediated by DLPFC-NAcc FC), a potential brain biomarker that could be an intervention target. These findings provide a compelling case to explore whether this brain biomarker can be modulated to enhance patients' ability to remain abstinent. Based on the above literature, there is a need to investigate non-invasive methods that can be used to increase FC between DLPFC and NAcc both in stimulant use disorder and alcohol use disorder. Because stimulant use and alcohol use are a very common incidence in the USA and both are a high burden on society, the current protocol will recruit both individuals with alcohol and stimulant use disorder.

Existing Literature: Executive functioning, the ability to change maladaptive behavior, depends on DLPFC input to NAcc (Gruber, Hussain, & O'Donnell, 2009). DLPFC transmits reward representations to NAcc through glutamatergic projections that guide goal-directed behavior (Ballard & Knutson, 2009). If DLPFC fails to activate when required, a common observation in substance use disorder, target neurons in the NAcc core do not receive critical information needed to select the appropriate outcome, causing acquired maladaptive response patterns to persist (e.g. drug consumption) (Gruber et al., 2009). Higher FC between DLPFC and NAcc may be achieved by stimulating DLPFC while subjects perform engaging executive functioning tasks. Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that can modulate brain connectivity. DLPFC stimulation may increase input to NAcc to facilitate proper selection of goal-directed behavior and may also decrease craving in individuals with substance use disorder (Boggio et al., 2008). Genetics and treatment response: A source of treatment response variability could stem from differences between participants in baseline genetic profiles or epigenetic changes over the course of treatment. Genetic polymorphisms, especially in genes important for neuroplasticity, may also mediate neuroplastic changes underlying the effects of tDCS (Chhabra et al., 2016), as has been demonstrated with gene BDNF (Antal et al., 2010; Fritsch et al., 2010). In light of these genetic influences on key tenants of our study - i.e. treatment response in alcohol use disorder and physiological effects of tDCS - we will collect genetic samples from participants to determine whether genetic or epigenetic variations may affect response to the cognitive training and tDCS intervention. This information may help inform the development of more individually-tailored treatment protocols in the future. As this is a secondary aim, participants will be given the choice in the Consent Form to opt in or out of the genetic sampling procedure.

Primary Endpoint/Event/Outcome: In a double-blind randomized design, 80 abstinent (3 weeks abstinent) individuals, 40 with Alcohol Use Disorder (AUD) and 40 with Stimulant Use Disorder (SUD) recruited from addiction treatment facilities will receive 10 sessions of either (i) transcranial direct current stimulation (tDCS) to PFC or (ii) sham-tDCS. All subjects will perform executive functioning tasks during each tDCS intervention (active or sham) to prime the engagement of the NAcc-PFC brain circuit. We have unpublished preliminary data indicating that the additional 5 treatment sessions (10 vs. 5) will likely improve outcomes and result in larger effect sizes. Follow-up interviews will be conducted monthly out to 4 months post intervention cessation (exact timepoint depending on participant availability) to query relapse status. We are expanding follow up visits out to 4 months because we have reason to believe that treatment effects could last up to 6 months post treatment. Tracking outcomes out to 4 months will be necessary to demonstrate durability of treatment benefits. Dependent variables will be (i) change in cognitive performance between pre- and post-intervention, and (ii) relapse status after study participation. The Specific Aims are to determine if the intervention: (A1) is feasible and safe in individuals with SUD and AUD, (A2) induces cognitive performance changes, and (A3) is related to relapse status in the months following study completion. A fourth exploratory aim is to examine relationships between genetic variants, epigenetic changes and (A2-3).

To evaluate feasibility (A1), withdrawal and retention policies are described in Section 12.0. To evaluate safety (A1), we will use the Treatment Side Effects Questionnaire to record intervention side effects. Based on our previous alcohol tDCS study and studies from other research groups, we hypothesize that the intervention will be feasible and safe.

To evaluate cognitive performance changes (A2), we will compare cognitive performance change from pre-intervention to post-intervention) between active tDCS and sham groups. We hypothesize that the active tDCS group will have a larger improvement in cognitive performance than the sham group.

To evaluate relapse status at all monthly follow-up visits, we will administer the Timeline Follow Back (Sobell and Sobell 1996), questionnaire and saliva/urine samples at each follow-up. Based on our alcohol pilot study and literature on the effects of tDCS in other addictions (Lupi et al. 2017; Batista et al. 2015), we hypothesize that the active tDCS group will have lower relapse rates and longer abstinence periods than the sham group.

Secondary Endpoint(s)/Event(s)/Outcome(s): To determine generalization and durability of cognitive training, patients will be asked to complete the following tasks at pre-intervention, post-intervention, and at 2 monthly follow up visits to examine generalization and durability effects of training: D-KEFS Trail Making Test, D-KEFS Verbal Fluency, D-KEFS Color Word, Digit-Span (WAIS), and Digit Symbol (WAIS).

ELIGIBILITY:
Inclusion Criteria:

* Abstinent from any substance or alcohol use (excluding caffeine or nicotine) for a minimum of 3 weeks at study enrollment
* Has the intention to remain in their treatment program(s) until the end of the intervention portion of the study.
* Able to provide written consent and comply with study procedures.
* Meets the MINI 7 diagnostic criteria for either stimulant use disorder (SUD) or alcohol use disorder (AUD).

Exclusion Criteria:

* Any medical condition or treatment with neurological sequelae (i.e. stroke, tumor, HIV)
* Over 9 months of abstinence from substance use
* A head injury resulting in a loss of consciousness exceeding 30 minutes (i.e., moderate or severe TBI)
* Presence of a condition that would render study measures difficult or impossible to administer or interpret
* Age outside the range of 18 to 65
* Primary current substance use disorder diagnosis (according to MINI 7 diagnostic criteria) for a substance other than stimulant or alcohol, except for caffeine or nicotine (Nicotine use will be recorded but is not exclusionary)
* Entrance to the treatment program under a court mandate. (i.e. legally incarcerated)
* History of ECT or cortical energy exposure within the past 6 months, including participation in any other neuromodulation studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Percent of participants with clean drug screens | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Kelvin Lim, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Fairview, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT04426214/ICF_000.pdf